CLINICAL TRIAL: NCT02023320
Title: A Randomized, Double-blind, Parallel Group Study to Evaluate the Effect of Blueberry Dry Powder on Prediabetes
Brief Title: Effects of Blueberry Dry Powder on Glycemic Status in Subjects With Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Agricultural Producers' Cooperative Corporation Shinpo-en (Unknown)
Responsible Party: Principal Investigator, Fumiko Higashikawa, Associate Professor, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: eki-842
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose of blueberry dry powder (Experimental): 0.5 g blueberry dry powder, twice a day for 12 weeks
  Interventions: Dietary Supplement: Low dose of blueberry dry powder
- High dose of blueberry dry powder (Experimental): 5.0 g blueberry dry powder, twice a day for 12 weeks
  Interventions: Dietary Supplement: High dose of blueberry dry powder

INTERVENTIONS:
Dietary Supplement: Low dose of blueberry dry powder
  Arms: Low dose of blueberry dry powder
Dietary Supplement: High dose of blueberry dry powder
  Arms: High dose of blueberry dry powder

SUMMARY:
The purpose of the present study is to evaluate the effect of blueberry dry powder on glycemic status (fasting plasma glucose, 2h glucose concentration after the oral glucose tolerance test (OGTT), or HbA1c) in subjects with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose 110-125 mg/dL

Exclusion Criteria:

* Taking anti-diabetic drugs
* Taking drugs or functional food that may affect blood glucose level
* Fruit allergy
* Pregnant or nursing a child
* Participation in any clinical trial within 90 days of the commencement of the trial
* Renal or hepatic dysfunction
* Heart disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in fasting plasma glucose from baseline | Every 6 weeks (Overall 12 weeks)
Change in 2h glucose concentration after the oral glucose tolerance test (OGTT) from baseline | Weeks 0 and 12
Change in HbA1c from baseline | Weeks 0 and 12

SECONDARY OUTCOMES:
Change in glycoalbumin from baseline | Every 6 weeks (Overall 12 weeks)
Change in fasting insulin from baseline | Weeks 0 and 12
Change in homeostasis model assessment-insulin resistance (HOMA-R) from baseline | Weeks 0 and 12
  HOMA-R is calculated as fasting insulin (mU/mL) x fasting glucose (mg/dL) / 405
Change in serum C-peptide from baseline | Weeks 0 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Fumiko Higashikawa, PhD, Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Hiroshima, Japan